CLINICAL TRIAL: NCT05120830
Title: Phase 1/2 Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of NTLA-2002 in Adults With Hereditary Angioedema (HAE)
Brief Title: NTLA-2002 in Adults With Hereditary Angioedema (HAE)
Acronym: NTLA-2002
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ITL-2002-CL-001
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Phase 1 is an open label non-randomized study Phase 2 is a randomized, double-blind, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 Study Arm (Experimental): Participants assigned to 1 of 3 dose-escalation cohorts will receive a single dose of NTLA-2002 on Day 1 and will then be followed for 104 weeks. Primary observation period is 16 weeks.
  Interventions: Biological: Biological NTLA-2002
- Phase 2 Experimental Study Arm (Experimental): Participants randomized to NTLA-2002 (2 dose levels), will receive a single dose of NTLA-2002 on Day 1 and will then be followed for 104 weeks. Primary observation period is 16 weeks.
  Interventions: Biological: Biological NTLA-2002
- Phase 2 Placebo Comparator Study Arm (Placebo Comparator): Participants randomized to placebo will receive IV normal saline on Day 1 and will then be followed for up to 104 weeks. Primary observation period is 16 weeks.
  Interventions: Other: Normal Saline IV Administration
- Placebo Crossover and Follow-On Dosing Substudy Arm (Experimental): Participants assigned to this Substudy Arm (participants who previously received either 25mg or placebo only) will have the opportunity to receive a single dose of NTLA-2002 (50mg) and will then be followed for 52 weeks.
  Interventions: Biological: Biological NTLA-2002

INTERVENTIONS:
Biological: Biological NTLA-2002 — CRISPR/Cas9 gene editing system delivered by LNP for IV administration
  Arms: Phase 1 Study Arm; Phase 2 Experimental Study Arm; Placebo Crossover and Follow-On Dosing Substudy Arm
Other: Normal Saline IV Administration — The administration of IV normal saline
  Arms: Phase 2 Placebo Comparator Study Arm

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, activity, pharmacokinetics, and pharmacodynamics of NTLA-2002 in adults with Hereditary Angioedema (HAE).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Diagnosis of HAE Types I or II
3. Ability to provide evidence of HAE attacks to meet the screening requirement
4. Subjects must have access to, and the ability to use, ≥ 1 acute medication(s) to treat angioedema attacks.
5. Adequate chemistry and hematology measures at screening
6. Subjects must agree not to participate in another interventional study for the duration of this trial.
7. Subjects must be capable of providing signed informed consent

Exclusion Criteria:

1. Concurrent diagnosis of any other type of recurrent angioedema
2. Subjects who have known negative reaction or hypersensitivity to any lipid nanoparticles (LNP) component.
3. Any condition that, in the Investigator's opinion, could adversely affect the safety of the subject.
4. Unwilling to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of NTLA-2002 as determined by adverse events (AEs) and dose limiting toxicities (DLTs) | From NTLA-2002 infusion up to week 104 post-infusion
  (Phase 1 only)
Number of HAE attacks per month (Weeks 1-16) | From study drug infusion up to week 16 post-infusion
  (Phase 2 only)

SECONDARY OUTCOMES:
Change from baseline in total plasma kallikrein protein level | From NTLA-2002 infusion up to week 104 post-infusion
  (Phase 1 & 2)
Plasma and urine concentrations for DMG-PEG2k, LP000001, Cas9 mRNA, and sgRNA | From NTLA-2002 infusion up to week 104 post-infusion
  (Phase 1 & 2)
Safety and tolerability of NTLA-2002 as determined by AEs | From study drug infusion up to week 104 post-infusion
  (Phase 2 only)
Number of HAE attacks per month (Weeks 5-16) | From week 6 post-infusion up to week 16 post-infusion
  (Phase 2 only)
Number of HAE attacks per month requiring acute therapy (Weeks 1-16, Weeks 5-16) | From study drug infusion up to week 16 post-infusion
  (Phase 2 only)

CONTACTS AND LOCATIONS:
Locations (9):
- Clinical Trial Site, Campbelltown, Australia
- France (3):
  - Clinical Trial Site, Grenoble
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Paris
- Germany (2):
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Frankfurt
- Clinical Trial Site, Amsterdam, Netherlands
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cohn DM, Gurugama P, Magerl M, Katelaris CH, Launay D, Bouillet L, Petersen RS, Lindsay K, Aygoren-Pursun E, Maag D, Butler JS, Shah MY, Golden A, Xu Y, Abdelhady AM, Lebwohl D, Longhurst HJ. CRISPR-Based Therapy for Hereditary Angioedema. N Engl J Med. 2025 Jan 30;392(5):458-467. doi: 10.1056/NEJMoa2405734. Epub 2024 Oct 24. PMID 39445704
- [Derived] Longhurst HJ, Lindsay K, Petersen RS, Fijen LM, Gurugama P, Maag D, Butler JS, Shah MY, Golden A, Xu Y, Boiselle C, Vogel JD, Abdelhady AM, Maitland ML, McKee MD, Seitzer J, Han BW, Soukamneuth S, Leonard J, Sepp-Lorenzino L, Clark ED, Lebwohl D, Cohn DM. CRISPR-Cas9 In Vivo Gene Editing of KLKB1 for Hereditary Angioedema. N Engl J Med. 2024 Feb 1;390(5):432-441. doi: 10.1056/NEJMoa2309149. PMID 38294975